CLINICAL TRIAL: NCT03429348
Title: Evaluation of Post-Exposure Sauna Treatment of Firefighters - A Pilot Study, Institutional Review Board# 1801201082
Brief Title: Evaluation of Post-Exposure Sauna Treatment of Firefighters - A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1801201082
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Results first posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2019-04

CONDITIONS: Post-fire Rehabilitation of Firefighters in Sauna
Keywords: Firefighter; Post-Fire Rehabilitation; Sauna

STUDY DESIGN:
Intervention Model Description: Working with firefighters during training fire exercises, Dr. Jeff Burgess and his study team will compare a chemical commonly excreted in firefighter urine samples after firefighting to assess the value of adding sauna to rehab post-fire. Firefighter heart rate and temperature will be monitored using a core body temperature/heart rate monitor data recorder. Urine will be collected for 12 hours immediately before the scheduled training fire and for 12 hours afterwards. After the fire, the firefighter will perform the standard rehab. During this time, the University of Arizona (UA) study team will randomly select half of the firefighters to an additional sauna rehab and the other half of the firefighters to no additional rehab. Dermal (skin) wipe samples will be taken off the calf, arm, and neck before the fire, before standard rehab, and after sauna/no additional treatment. A post-fire survey will be administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No additional rehabilitation (No Intervention): No additional rehabilitation will be done
- Sauna rehabilitation (Other): An additional rehabilitation in a sauna will be done
  Interventions: Other: Sauna Rehabilitation

INTERVENTIONS:
Other: Sauna Rehabilitation — Firefighters selected for sauna rehabilitation will spend time in a sauna
  Arms: Sauna rehabilitation

SUMMARY:
Firefighters are at increased risk of cancer, and both inhalation and dermal routes contribute to overall exposure to carcinogens, including polycyclic aromatic hydrocarbons (PAHs). The purpose of the current study is to determine if post-fire firefighter rehabilitation in an infrared sauna: a) affects absorption of PAHs as measured by urinary metabolites; and b) changes core body temperature and heart rate.

DETAILED DESCRIPTION:
An initial four firefighters will be evaluated for change in PAHs associated with standard fire department flashover training to determine if urinary PAH metabolites increase following exposure, comparing baseline urine samples (collected for up to 12 hours before the training fire) to a repeat urine sample (collected up to 12 hours after cessation of the training fire.) If a significant increase is not seen, then repeat testing with four firefighters will be completed using burn room training scenarios. Air monitoring during the training periods may be carried out with standard industrial hygiene instruments.

Stage 2: Once a significant increase in PAHs has been documented, the associated training scenario (flashover training or alternate live fire training), testing will be carried out in 20 subjects. Prior to starting the training scenario, the firefighters will provide a urine sample (collected over a time period of 12 hours prior to the training fire), swallow a core temperature probe and wear a monitor for recording both their core temperature and heart rate. In addition, dermal wipes will be collected prior to the training fire. Air monitoring during the training periods will be carried out with standard industrial hygiene instruments. Following cessation of the training scenario, the subjects will follow their standard fire department procedures, which may involve using skin wipes and showering. The subjects will then be randomized to either an infrared sauna treatment, with or without exercising as determined by the fire department protocol, or no additional treatment, following their fire department protocols. Repeat dermal wipes will be collected in all subjects. Core temperature and heart rate will be monitored for up to 8 hours after training scenario. The subjects will collect all their urine after the fire training for a period of 12 hours. The urine will be analyzed for urinary PAH metabolites and potentially other toxicants from the fire, and, dependent on the available budget, similar evaluations may be carried out on the skin wipes.

ELIGIBILITY:
Inclusion Criteria:

* Are employed as an active fire responder by the Fire Department
* Are scheduled for a training fire exercise by the Fire Department in the next year
* Are currently a non-smoker (including cigarettes, cigars and e-cigarettes)
* Cannot have any contraindications to the core temp pill, which are:

  * weight less than 80 pounds
  * known or suspected obstructive disease of GI tract, including but not limited to diverticulitis and inflammatory bowel disease
  * exhibit or have a history of disorders or impairment of the gag reflex
  * have had a previous gastrointestinal surgery
  * have any diseases or disorders of the esophagus
  * will be undergoing Nuclear Magnetic Resonance (NMR) or MRI scanning less than 3 days after swallowing the sensor
  * have a low motility disorder of the gastrointestinal tract including but not limited to ileus
  * have a cardiac pacemaker or other implanted electromedical device
  * have a swallowing disorder

Exclusion Criteria:

* Are NOT employed as an active fire responder by the Fire Department
* Are NOT scheduled for a training fire exercise by the Fire Department in the next year
* Are currently a smoker (including cigarettes, cigars and e-cigarettes)
* Has one of the contraindications to the core temp pill

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jefferey L Burgess, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crinnion W. Components of practical clinical detox programs--sauna as a therapeutic tool. Altern Ther Health Med. 2007 Mar-Apr;13(2):S154-6. PMID 17405694
- See also: Use of the Hubbard Sauna Detoxification Regimen to Improve the Health Status of New York City Rescue Workers Exposed to Toxicants — http://www.getdetoxinated.com/docs/townsend_letter-04-2006.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Additional Rehabilitation | Sauna Rehabilitation
Started | 12 (4 participants had no additional rehab & had no corresponding sauna rehab participant to compare to.) | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Additional Rehabilitation | Sauna Rehabilitation | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 12 | 20
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Urinary PAH-OHs [Mean (Standard Deviation); unit: ng/L] | 10364.2 (2.7) | 6964.1 (1.7) | 8495.7 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Urinary Excretion of Hydroxylated PAHs (PAH-OHs)
Description: Urine samples from firefighters post-fire will be measured for hydroxylated PAHs (PAH-OHs) and the concentration compared to pre-fire urine concentrations of PAH-OHs
Time Frame: 12 hours for urine collection
Measure: Mean (Standard Deviation); unit: ng/L
Groups:
- Baseline No Additional Rehabilitation Group Urine PAH-OH Sum: Urine samples were analyzed for PAH-OHs The derivatized extracts were analyzed with gas chromatography mass spectroscopy (GC-MS). The sum of the PAH-OHs was determined for the baseline control group samples.
- Post-fire No Additional Rehabilitation Group: Urine samples were analyzed for PAH-OHs The derivatized extracts were analyzed on a GC-MS. The sum of the PAH-OHs was determined for the post-fire samples for the control group.
- Baseline Sauna Rehabilitation Group Urine PAH-OH Sum: Urine samples were analyzed for PAH-OHs The derivatized extracts were analyzed on a GC-MS. The sum of the PAH-OHs was determined for the baseline sauna group.
- Post-fire Sauna Rehabilitation Group: Urine samples were analyzed for PAH-OHs The derivatized extracts were analyzed on a GC-MS. The sum of the PAH-OHs was determined for the post-fire sauna group.
Arm/Group | Baseline No Additional Rehabilitation Group Urine PAH-OH Sum | Post-fire No Additional Rehabilitation Group | Baseline Sauna Rehabilitation Group Urine PAH-OH Sum | Post-fire Sauna Rehabilitation Group
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng/L | 10364.2 (2.7) | 40012.1 (2.6) | 6964.1 (1.7) | 22604.3 (1.6)
Statistical Analysis 1: Comparison: Baseline Sauna Rehabilitation Group Urine PAH-OH Sum vs Post-fire Sauna Rehabilitation Group; Test type: Superiority; p = 0.0000009, t-test, 2 sided; We are comparing the log transformed values; Mean Difference (Final Values) = 1.18
Statistical Analysis 2: Comparison: Baseline No Additional Rehabilitation Group Urine PAH-OH Sum vs Post-fire No Additional Rehabilitation Group; Test type: Superiority; p = 0.000018, t-test, 2 sided; We are comparing the log transformed values; Mean Difference (Final Values) = 1.35

ADVERSE EVENTS:
Time Frame: Subjects were monitored for 12 hours following completion of their live-fire burn training exercise.
Description: Following the live-fire exercises, all firefighters were monitoring for heart rate and blood pressure. No one was allowed to leave the rehabilitation station until these parameters met the fire department protocols. The firefighters brought urine back to the researchers at 12 hours following cessation of their training exercise. While we did not specifically collect data on deaths or serious adverse events at 12 hours, at that time none were reported.
Arm/Group | No Additional Rehabilitation | Sauna Rehabilitation
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
This study involved idealized treatment conditions which included shorter intervals between exiting the fire and entry into the sauna than could likely be achieved with actual structure fires.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT03429348/Prot_000.pdf